CLINICAL TRIAL: NCT04983342
Title: Apollo Device for Fatigue in Metastatic Breast Cancer
Brief Title: Apollo Device for Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margaret Quinn Rosenzweig (Other)
Collaborators: Apollo Neuroscience, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Margaret Quinn Rosenzweig, Distinguished Service Professor of Nursing, Professor of Medicine Director of Catchment Area Research - Hillman Cancer Center, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCC 20-243
Record Dates: First submitted 2021-07-15; First posted 2021-07-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Fatigue; Metastatic Breast Carcinoma
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm pilot design -pre and post
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apollo Armband (Experimental): Armband that can be worn on the ankle, wrist, or arm with two adjustable fabric straps. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy, combatting fatigue and pain.
  Interventions: Device: Apollo Armband

INTERVENTIONS:
Device: Apollo Armband — The Apollo armband is approximately the size of an Apple Watch and can be worn on the ankle, wrist, or arm with two adjustable fabric straps. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy, combatting fatigue and pain. In addition to the wearable, Apollo is a software system that curates music for the body, rather than for the ears.

SUMMARY:
This is a single-arm, open label pilot intervention study with outcomes measured by electronic survey and chart review evaluating a wearable device called Apollo, which is similar to a FitBit but emits vibrations. Our primary objective is to assess whether or not Apollo can help with symptoms of fatigue and pain in patients with Metastatic Breast Cancer (MBC).

DETAILED DESCRIPTION:
This study aims to provide preliminary data on the efficacy and tolerability of the Apollo device in the management of fatigue and pain in patients with Metastatic Breast Cancer (MBC).

Apollo is about the size of an Apple Watchand can be worn on the ankle, wrist, or armwith two adjustable fabric straps. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy. In addition to the wearable, Apollo is a software system that curates music for the body, rather than for the ears. The scientific principles guiding the use of Apollo and mechanistic understanding of its effects on the body are consistent with the understanding of how music and therapeutic touch effect the body to convey feelings of energy, focus, or relaxation by sending safety signals to the emotional cortex (limbic system) in the brain. Similar to music and touch used to facilitate a healing response in the body, there are no known side effects to this type of therapy.

The PROMIS-Fatigue scale and the Functional Assessment of Cancer Therapy Fatigue (FACT-F) are instruments that have been previously validated in multiple diseases and will be used in this study. Preliminary data on indices of pain, use of PRN pain medications, health-related quality of life, sleep, anxiety and depression and tolerability/frequency of use with the Apollo device in MBC will also be evaluated using:

* PROMIS pain scale
* Use of pain medications
* Health-related quality of life (HRQOL) using PROMIS-29
* PROMIS Sleep
* Hospital Anxiety and Depression Scale (HADS)
* Usage data from Apollo app

This study aims to identify improvement of fatigue symptoms from baseline after 4 and 8 weeks of Apollo use. Improvements in pain, quality of life, use of PRN pain medication, anxiety and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer diagnosis
* Fatigue score of 4 or greater at last clinic visit

Exclusion Criteria:

* Not able to read and understand English
* Use of Beta Blockers,
* Use of medications for serious mental illness

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most MBC is among females - males are excluded due to lack of generalizability
Enrollment: 27 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue (PROMIS-Fatigue) | Up to 8 weeks
  Change from baseline to 4 and then 8 weeks as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue scale, which measures the presence of fatigue and its interference with life. PROMIS-Fatigue includes 6 items with scores 1-5 for each item, total scores 6-30. Lower scores indicate less fatigue and interference from fatigue.
Change in Fatigue (FACT-F) | Up to 8 weeks
  Change from baseline to 4 and then 8 weeks as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 40-item, 5 choice/item measure ranging from 0 (Not at all) to 4 (Very much) that assesses self-reported fatigue and its impact upon daily activities and function, 0-160 is the total score with higher scores indicating better QOL, the lower the fatigue symptoms. The recall period refers to the "past 7 days".

SECONDARY OUTCOMES:
Degree of Pain | Up to 8 weeks
  The PROMIS Pain scale will be used to measure the degree of pain experienced. PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health. The Pain Intensity part is a 3-item scale focuses on representing the full range of possible pain intensity using psychometric properties and clinical input, with frequency (never to always) and severity (none to very severe) Likert-type response scales. The final measure includes three items rating pain from "Had no pain" = 1 to "Very severe" = 5. Scores range from 3-15, with higher scores indicating more severe pain. The pain interference part consists of 6 items ranging 1 through 5 - total scores 6-30. Higher scores indicate higher degrees of interference with important aspects of life. The recall period for all pain quality items is the past 7 days.
Use of pain medications | Up to 8 weeks
  The dosage of specific medications will be recorded.
Health Related quality of life (HRQOL) | Up to 8 weeks
  Quality of Life will be assessed using the the Promis-29. The Promis-29 is a short form assessment containing four items from each of seven PROMIS domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) plus one pain intensity question (0-5 numeric rating scale). Higher scores indicate greater difficulty and/or poorer quality of life.
Promis Sleep Measurement | Up to 8 weeks
  Measure of sleep difficulty by first asking the participant to rate their sleep quality (very poor, poor, fair, good, very good). Participants are then ask to rate their sleep as, "refreshing; had a problem with sleep; had difficulty falling asleep; sleep was restless, hard to get to sleep, worried about not being able to get to sleep, unsatisfied with their sleep. Response scale: Not at all, A little bit, Somewhat, Quite a bit, Very much. Scoring scale is 1-5 (Very poor ,poor, fair, good, very good) Total scores range from 8-45, with higher numbers indicating better sleep.
Hospital Anxiety and Depression Scale (HADS) | Up to 8 weeks
  Hospital Anxiety and Depression Scale (HADS) assesses both anxiety and depression, focusing on non-physical symptoms so that it can be used to diagnose depression in people with significant physical ill-health. Self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). The maximum score is therefore 21 for depression and 21 for anxiety. A score of 11 or higher indicates the probable presence of the mood disorder with a score of 8 to 10 being just suggestive of the presence of the respective state. The HADS questionnaire takes 2-5 min to complete and is comprised of seven questions for anxiety and seven questions for depression, with anxiety and depression questions interspersed within.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Q Rosenzweig, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
If investigators want to see de-identified data we will work with Apollo company to share data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months following last patient accrual.